CLINICAL TRIAL: NCT04483219
Title: A Single-arm, Multicenter Phase II Clinical Study to Evaluate the Efficacy and Safety of Tyrosine Kinase Inhibitor (TKI) in Combination With Anti-PD-1 Antibody in TKI-responded Microsatellite Stability/Proficient Mismatch Repair (MSS/pMMR) Metastatic Colorectal Adenocarcinoma.
Brief Title: Tyrosine Kinase Inhibitor (TKI) + Anti-PD-1 Antibody in TKI-responded Microsatellite Stability/Proficient Mismatch Repair (MSS/pMMR) Metastatic Colorectal Adenocarcinoma.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Medical University, China (Other)
Responsible Party: Principal Investigator, Jingdong Zhang, Director, China Medical University, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TRAP
Record Dates: First submitted 2020-07-14; First posted 2020-07-23 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-09

CONDITIONS: MSS; pMMR; Metastatic Colorectal Adenocarcinoma
Keywords: tyrosine kinase inhibitors (TKIs); programmed cell death protein 1 (PD-1); microsatellite stable/proficient mismatch repair (MSS/pMMR); metastatic colorectal adenocarcinoma (mCRC); trial
MeSH Terms: conditions — Parkinson Disease 4, Autosomal Dominant Lewy Body

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TKI ± anti-PD-1 antibody (Experimental): According to response to TKI, the combination of anti-PD-1 treatment would be determined.
  Interventions: Drug: TKI ± anti-PD-1 antibody

INTERVENTIONS:
Drug: TKI ± anti-PD-1 antibody — After one cycle of TKI, evaluations would be performed according to RECIST v 1.1. (1) obvious response (A): CR, PR or shrunken SD, or cavitation in metastatic lung lesions, or decrease in the density of liver metastatic targets ≥15%; (2) general response (B): enlarged SD; (3) poor response (C): PD. TKI ＋ anti-PD-1 antibody will be administered in group A. The subjects in group C will exit the study. The subjects in group B will continue TKI for another one cycle, the obvious response subjects will entered group A, the general response subjects will keep in arm B and continue the TKI monotherapy, and the poor response subjects will exit the study.
  1. Fruquintinib 5mg or regorafenib 120mg, qd po, 3 weeks, Q4w. (The investigators decide to choose fruquintinib or regorafenib)
  2. Toripalimab injection 240mg, Q3w, until the disease progresses or lasts for two years.

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of fruquintinib or regorafenib in combination with anti-PD-1 antibody in TKI (fruquintinib or regorafenib)-responded MSS/pMMR metastatic colorectal adenocarcinoma.

DETAILED DESCRIPTION:
At present, the later-line treatment of metastatic colorectal cancer (mCRC) can bring benefits to subjects. However, the overall efficacy of treatment is still low. The programmed cell death protein 1 (PD-1) blockade alone in MSS/pMMR mCRC is inefficiency, highlighting a need for strategies that converse the immunity suppressive to immunity supportive microenvironment. Fruquintinib and regorafenib are multi-target TKI mainly for angiogenesis, which has the following characteristics: cause tumor necrosis and release a lot of new antigens, improve the microenvironment of immunosuppression, and induce tumor vascular normalization. In addition to killing tumor cells, fruquintinib and regorafenib could also converse the immunity suppressive to immunity supportive microenvironment, which could sensitize PD-1 blockade, ultimately improve the prognosis of patients with MSS/pMMR mCRC.

This prospective study is a single-arm, multicenter phase II clinical study to evaluate the efficacy and safety of fruquintinib or regorafenib in combination with anti-PD-1 antibody in TKI (fruquintinib or regorafenib)-responded MSS/pMMR metastatic colorectal cancer.

In this prospective study, the 9-month PFS rate in subjects receiving TKI followed by TKI in combination with anti-PD-1 antibody, will be used as primary outcome measures and 53 subjects will be recruited.

After fully informed and signed the informed consent, the subjects will receive one cycle of TKI (fruquintinib or regorafenib) treatment after enrollment. According to response to TKI, the subjects will be divided into three arms. The definition of response to TKI are as follows: (1) obvious response to TKI (arm A)：effective imaging changes, including reduction of target lesion diameter to CR, PR or shrunken SD (based on response evaluation criteria in solid tumors, RECIST v 1.1), or cavitation in metastatic lung lesions, or decrease in the density of liver metastatic target lesions ≥15%; (2) general response to TKI (arm B): enlarged SD (based on RECIST v 1.1); (3) poor response to TKI (arm C): PD (based on RECIST v 1.1). TKI in combination with anti-PD-1 antibody will be administered in arm A. The subjects in arm C will exit the study. The subjects in arm B will continue to take TKI for another one cycle. After that, the obvious response subjects will be entered group A, the general response subjects will keep in arm B and continue the TKI monotherapy, and the poor response subjects will exit the study. The administration of arm A or B will be last until disease progression or intolerable toxicity，anti-PD-1 antibody can be applied for up to 2 years.

The first two imaging evaluations would be performed every 4 weeks after the beginning of treatment to evaluate TKI response, and then once every 6 weeks, until the end of treatment, withdrawal of informed consent or death. The TKI response would be assessed according to RECIST v1.1 criteria and effective imaging changes (cavitation in metastatic lung lesions, or decrease in the density of liver metastatic target lesions ≥15%). The efficacy of TKI followed by TKI in combination with anti-PD-1 antibody would be evaluated based on immune-related RECIST (iRECIST) v1.1 criteria.

PD-1/PD-L1 expression, T lymphocyte infiltration, T lymphocyte subsets in peripheral blood, granulocyte to lymphocyte ratio, tumor mutant burden (TMB), circulating tumor DNA (ctDNA), exosomes，etc.，will be measured and monitored during the treatment. In addition，the safety evaluation will be carried out according to the standard of adverse reaction classification (Common Terminology Criteria for Adverse Events, CTCAE v5.0)

ELIGIBILITY:
Inclusion Criteria:

* Subjects who voluntarily participated in the study, signed the written informed consent form, and could comply with the protocol of study.
* Male or female of age 18-75 years.
* Subjects with colorectal adenocarcinoma who were histopathologically confirmed, and with locally advanced (unresectable) or mCRC.
* Subjects who underwent standard antitumor therapies (fluorouracil, oxaliplatin, irinotecan were used, with or without administration of bevacizumab and/or cetuximab).
* Patients with MSS/pMMR mCRC (immunohistochemistry, polymerase chain reaction or next-generation sequencing can be used).
* All adverse reactions associated with drug use or surgery were reduced to grade 0-1 (according to Common Terminology Criteria for Adverse Events (CTCAE) version 5.0) or to a level required by the protocol criteria.
* The presence of at least one measurable lesion by computed tomography (CT) or magnetic resonance imaging (MRI).
* Eastern Cooperative Oncology Group (ECOG) performance status score of ≤ 1.
* Subjects with life expectancy ≥ 12 weeks.
* Adequate important organs functions: bone marrow function (neutrophil count ≥ 1.5×10^9/L; platelet ≥ 80×10^9/L; hemoglobin ≥ 90 g/L), liver function (serum albumin ≥ 28 g/L; total bilirubin ≤ 1.5×upper limit of normal (ULN); alanine aminotransferase and aspartate aminotransferase ≤ 3×ULN, or ≤ 5×ULN if liver metastases are present), renal function (serum creatinine ≤ 1.5×ULN or creatinine clearance (CrCl) ≥ 40 mL/min, using the Cockcroft-Gault formula; urine protein < 2+; 24h urinary protein content < 1.0 g/24h if urinary protein ≥ 2+ ), coagulation function (international normalized ratio or activated partial thromboplastin time ≤ 2×ULN), thyroid function (thyrotropin ≤ 1×ULN).

Exclusion Criteria:

* Known microsatellite instability high (MSI-H) mCRC.
* Participation in another study with intervention or drugs within the past 4 weeks.
* Performing surgery and incomplete recovery within the past 4 weeks.
* Subjects with active autoimmune diseases or with related history. Subjects with controlled type I diabetes or hypothyroidism with substitution therapy may be included for further screening.
* Any conditions requiring corticosteroids (> 10 mg per day of prednisone or equivalent) or immunosuppressive drugs as systemic treatment within the past 1 week.
* Other active malignancy within the past 5 years, except for the cured limited cancer (such as basal cell carcinoma, carcinoma in situ of the prostate or cervix, etc.).
* Subjects with history of hepatic encephalopathy or confirmed metastases to central nervous system.
* Subjects with non-infectious pneumonia under steroid treatment within the past 6 months.
* Suffering from chronic or active infections, fever (≥ 38.5℃) within the past 1 week, or white blood cell count > 15×10^9/L), requiring systemic anti-infective treatment at the screening period, except for viral hepatitis.
* Subjects with any other abnormal condition that is inconsistent with the study medication, or may increase the risk of the subject，according to investigators' judgment.
* Congenital or acquired immunodeficiency (such as human immunodeficiency virus).
* Subjects with active hepatitis B virus (HBV) (HBV surface antigen positive and HBV-DNA > 2000 IU/ml) or hepatitis C virus (HCV) (HCV antibody and HCV-RNA positive).
* Subject who received a live attenuated vaccine within the past 4 weeks, or vaccination is planned during anti-PD-1 antibody treatment or within 5 months after the last treatment.
* More than mild pericardial effusion, massive pleural or/and peritoneal effusions need puncture and drainage at the screening period.
* Subjects with symptomatic heart and cerebrovascular diseases: heart failure (New York Heart Association class III or IV, left ventricular ejection fraction < 50%), uncontrolled hypertension or arrhythmias, serious cardiovascular and cerebrovascular events (acute coronary syndrome, stroke, thromboembolism, etc.) within the past 6 months.
* Known allergy to targeted drugs.
* Women being pregnant, or during lactation, or planning to get pregnant during the trial.
* Subjects with any other conditions judged by investigators would be excluded.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2020-07-24 (Actual); Primary Completion 2022-07-31 (Estimated); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
9-month progression-free survival (PFS) rate (in subjects receiving TKI followed by TKI in combination with anti-PD-1 antibody) | 9 months
  From the date of first dose of treatment to the first of either disease progression, relapse or death from any cause, evaluate patient PFS rate at 9 months

SECONDARY OUTCOMES:
Objective response rate (ORR) | 2 years
  Defined as the proportion of patients whose best overall response (BOR) is complete response (CR) or partial response (PR) assessed by iRECIST v1.1
Duration of response (DOR) | 2 years
  Defined as the time from CR or PR to disease progression or death.
Disease control rate (DCR) | 2 years
  Defined as the proportion of patients whose BOR is CR, PR, and stable disease (SD) assessed.
Progression-free survival (PFS) | 2 years
  Defined as the time from the date of the first dose of treatment to the date of the first documentation of disease progression or death, whichever occurs first.
Overall survival (OS) | 2 years
  Defined as the time from the date of the first dose of treatment until the date of death due to any cause.
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 2 years
  The grade of toxicity will be assessed using the NCI-CTCAE version 5.0.
Health-related quality of life (HRQOL) | 2 years
  Score according to quality of life scale.
Exploration of biomarkers | 2 years
  PD-1/PD-L1 expression, tumor-infiltrating lymphocytes, T lymphocyte subsets from peripheral blood samples, granulocyte-to-lymphocyte ratio, TMB, ctDNA, exosomes, dynamic changes in serum levels of protein tumor markers, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Jingdong Zhang, Principal Investigator — China Medical University, Liaoning Cancer Hospital & Institute,China
Locations (1):
- Cancer Hospital of China Medical University/Liaoning Cancer Hospital &Institute, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data will be available (including data dictionaries). All the individual participant data collected during the trial, after deidentification. All the study protocol, statistical analysis plan, informed consent form, clinical study report and analytic code will be available. The data will be available immediately following publication and no end date. The data will be shared with the researchers who provide a methodologically sound proposal to achieve aims in the approved proposal. The proposals should be directed to jdzhang@cancerhosp-ln-cmu.com.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Immediately following publication.No end date.
Access Criteria: Researchers who provide a methodologically sound proposal. The proposals should be directed to jdzhang@cancerhosp-ln-cmu.com.

REFERENCES:
- [Derived] Dong Q, Diao Y, Sun X, Zhou Y, Ran J, Zhang J. Evaluation of tyrosine kinase inhibitors combined with antiprogrammed cell death protein 1 antibody in tyrosine kinase inhibitor-responsive patients with microsatellite stable/proficient mismatch repair metastatic colorectal adenocarcinoma: protocol for open-label, single-arm trial. BMJ Open. 2022 Apr 4;12(4):e049992. doi: 10.1136/bmjopen-2021-049992. PMID 35379611